CLINICAL TRIAL: NCT01985984
Title: Outcome Prediction in Head&Neck Cancer Patients After Radiotherapy Using Multi-parameter Modelling: Disease Control, Toxicity and Quality of Life
Brief Title: Outcome Prediction in Head&Neck Cancer Patients After Radiotherapy
Acronym: OutcomeH&N
Status: Recruiting | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: 12-02-8/02-extern-6820
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Cancer
Keywords: Head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiation; Chemoradiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- H&N cancer patients: Patients with Head and Neck Cancer, treated with curative intent
  * Any tumor site
  * Stage I-IV, M0
  * Treated with radiotherapy alone or in combination with systemic therapy
  * Definitive radiotherapy or postoperative radiotherapy
  Interventions:
  * Radiation alone
  * Radiation in combination with systemic therapy
  Interventions: Radiation: Radiation alone; Radiation: Radiation in combination with systemic therapy

INTERVENTIONS:
Radiation: Radiation alone — Radiation alone
Radiation: Radiation in combination with systemic therapy — Radiation in combination with systemic therapy
  Other Names: Chemoradiation

SUMMARY:
The primary and general objective of the clinical introduction of the Standard Follow-up Program (SFP) as the current standard of care is to improve the quality of radiotherapy for head and neck cancer patients by reducing radiation-induced side effects without hampering treatment efficacy in terms of locoregional tumour control and overall survival and to systematically evaluate the beneficial effect of newly introduced radiation technology for this particular group of patients. The clinical introduction of the SFP will allow for a systematic and broad scale quality improvement cycle for head and neck cancer patients treated with radiotherapy. In fact, this methodology can be considered a kind of quality circle for the clinical introduction of new radiation techniques, aiming at continuous efforts for further improvement.

DETAILED DESCRIPTION:
For head and neck squamous cell carcinoma (HNSCC), radiation therapy is one of the mainstays of therapy either as definitive therapy alone or in combination with systemic therapy or following surgical resection as postoperative treatment. Nowadays there's great attention for personalized medicine which aims at offering a patient the treatment that best suits the individual patient and its tumor characteristics. To apply personalized therapy, we need accurate outcome prediction models for disease control, treatment related toxicity and quality of life.

The main factors used for predictive/prognostic nomograms are clinical factors, like patient-, tumor- and treatment related factors (1). Standard examples of these include age, gender, co-morbidity, smoking history, hemoglobin levels, tumor site, TNM stage, tumor volume, HPV-status, and others. For larynx cancer the nomogram was made publicly available on www.predictcancer.org.

However, we anticipate that other factors will contribute to the (improvement of) prediction models. These factors may include genomic analysis of tumor specimens, quantitative image analysis (radiomics), blood biomarkers, and/or tumor-tissue markers (2).

In addition, treatment-related parameters also need to be considered and these not only include factors like overall treatment time, use of systemic therapy, prescribed radiation dose and fraction dose. With new techniques using EPID dosimetry, it is now possible to measure the delivered radiation dose and compare this to the prescribed dose (3,4). This offers the potential to apply Dose Guide RadioTherapy (DGRT), which especially in HNSCC may have a large impact, because anatomical changes during fractionated therapy are known to occur and lead to dose changes to targets and organs at risk (5,6).

The final objective of this study is to integrate all potential prognostic factors and develop reliable nomograms both for tumor control as well as complications.

ELIGIBILITY:
Inclusion Criteria:

All patients planned for curatively intended primary or postoperative radiotherapy

Exclusion Criteria:

All patients planned for palliative radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Characteristics of the population:
  * Patients with Head and Neck Cancer, treated with curative intent
  * Any tumor site
  * Stage I-IV, M0
  * Treated with radiotherapy alone or in combination with systemic therapy
  * Definitive radiotherapy or postoperative radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-07; Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 years
  The overall survival will be calculated from the first day of treatment, either the first day of induction chemotherapy or the first day of radiotherapy in case of concomitant chemoradiation or radiation alone. An event is defined as death of any cause.

SECONDARY OUTCOMES:
disease free survival | 5 years
loco-regional control | 5 years
  Loco-regional control will be calculated from the first day of treatment, either the first day of induction chemotherapy or the first day of radiotherapy in case of concomitant chemoradiation or radiation alone. An event is defined as local recurrence and/or regional recurrence. These two events will be separately scored.

OTHER OUTCOMES:
Patient-rated symptoms and quality of life | 5 years
  quality of life (EORTC QLQ-C30, EORTC QLQ-H&N35, EuroQoL-EQ5D)
Acute and late toxicity scores, according to CTCv4.0 criteria | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: F Hoebers, MD, PhD, Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- Maastro Clinic, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No